CLINICAL TRIAL: NCT02511548
Title: Increasing Medical Male Circumcision Uptake in Orange Farm (South Africa): An Operational Study of Demand Creation
Brief Title: Increasing Medical Male Circumcision Uptake
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Progressus (Other)
Responsible Party: Principal Investigator, bertran Auvert, Scientific Investigator, Progressus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MCUptake
Record Dates: First submitted 2015-07-28; First posted 2015-07-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Circumcision, Male; Circumcision Status: Circumcised, Uncircumcised

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Financial incentive
  Interventions: Other: Financial incentive
- Control (No Intervention): No financial incentive

INTERVENTIONS:
Other: Financial incentive — Financial incentive will be proposed to participant of the intervention arm
  Arms: Intervention

SUMMARY:
The main objective of this study is to reach 80% circumcised men in a random sample of men living in the township of Orange Farm (South Africa).

DETAILED DESCRIPTION:
The World Health Organization and the United Nations Programme on HIV/AIDS recommend voluntary adult medical male circumcision as an intervention against HIV in Africa since 2007 and has estimated that achieving 80% male circumcision coverage would have a major public health impact. Despite evidence of its effectiveness, feasibility, cost-effectiveness and acceptability, its roll-out in Eastern and Southern Africa, the region where HIV prevalence is highest in the world, remains slow. Developing and testing innovative strategies to accelerate voluntary adult medical male circumcision roll-out is thus necessary. As a target community of this prevention method, Orange Farm (Gauteng Province) is a prime setting to conduct operational research. The team presenting this project conducted the first voluntary adult medical male circumcision randomized trial (ANRS-1265), successfully led the ANRS-12126 voluntary adult medical male circumcision roll-out, and has just completed the ANRS-12285 study on voluntary adult medical male circumcision and HIV incidence. Due to the roll-out, male circumcision prevalence increased from 12% in 2008 to 53% in 2011 in the township, but to date this prevalence has remained stagnant.

The main objective of this study is to reach 80% circumcised men in randomized clusters of Orange Farm (Gauteng Province), a township where voluntary adult medical male circumcision roll-out is ongoing since 2007.

Existing communication strategies will be revised and supplemented by personalised individual discussions to increase motivation for voluntary adult medical male circumcision and translate it into actual uptake.

The project consists of: 1) A preparatory phase to establish collaborations and prepare the communication activities, 2) a survey phase during which a) a mass communication campaign will be launched and b) 300 uncircumcised men selected from randomized clusters of Orange Farm will be recruited and undergo a baseline assessment including voluntary adult medical male circumcision general counselling, and 3) a follow-up phase during which repeated motivational interviews will be conducted to address their individual reasons for not being circumcised. Financial incentive will also be tested in a randomized trial.

Willing men will be referred to the free local voluntary adult medical male circumcision clinic and asked to attend an interview on the reasons that motivated them to become circumcised. At the end of the study, male circumcision prevalence among participants will be calculated. Factors associated with voluntary adult medical male circumcision uptake will be studied.

The survey phase will include a total of 600 uncircumcised and circumcised adult men. Among them, an expected 200 uncircumcised men will be included in the follow-up phase.

Participants will receive a financial compensation for their participation.

The study will last about 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Uncircumcised men
* Willing to participate
* Living in Orange Farm
* Able to speak and read English, Sotho or Zulu

Exclusion Criteria:

* Unable to give informed consent
* Planning to leave the study area within the next year

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2015-08; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Male circumcision uptake | 3 weeks
  The proportion of participants who will accept to become circumcised during the course of the study in each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Bertran Auvert, MD, PhD, Principal Investigator — University of Versailles

REFERENCES:
- [Background] Auvert B, Taljaard D, Rech D, Lissouba P, Singh B, Bouscaillou J, Peytavin G, Mahiane SG, Sitta R, Puren A, Lewis D. Association of the ANRS-12126 male circumcision project with HIV levels among men in a South African township: evaluation of effectiveness using cross-sectional surveys. PLoS Med. 2013;10(9):e1001509. doi: 10.1371/journal.pmed.1001509. Epub 2013 Sep 3. PMID 24019763
- [Background] Thirumurthy H, Masters SH, Rao S, Bronson MA, Lanham M, Omanga E, Evens E, Agot K. Effect of providing conditional economic compensation on uptake of voluntary medical male circumcision in Kenya: a randomized clinical trial. JAMA. 2014 Aug 20;312(7):703-11. doi: 10.1001/jama.2014.9087. PMID 25042290